CLINICAL TRIAL: NCT05666349
Title: Reirradiation (Re-RT) and Niraparib (NIRA) in Patients With Recurrent Glioblastoma (rGBM)
Brief Title: Reirradiation and Niraparib in Patients With Recurrent Glioblastoma
Acronym: RiNG
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funder support withdrawn 13-Oct-2023. Study did not open to recruitment.
Sponsor: University College, London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/142286; 2022-001706-22 (EudraCT Number)
Record Dates: First submitted 2022-11-02; First posted 2022-12-27 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Glioblastoma
Keywords: Niraparib; Glioblastoma; Re-irradiation
MeSH Terms: conditions — Glioblastoma | interventions — niraparib; Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niraparib and re-irradiation (re-RT) (Experimental): Patients will be treated with IMRT-based re-RT for a total dose of 35 Gy in 10 daily fractions over approx. 2 weeks. Patients will take niraparib daily from the first day of re-RT until documented progression or discontinuation due to unacceptable treatment-related toxicity or any other cause (whichever occurs sooner).
  Patients will be recruited in cohorts of 3. Following the completion of each dosing cohort and once the patients have completed the dose limiting toxicity (DLT) assessment window, the independent data monitoring committee (IDMC) will review the data for each patient. In conjunction with the statistical recommendations from the continual reassessment method (CRM), the IDMC will advise whether the dose for the next cohort should be escalated, de-escalated or stay at the current niraparib dose.
  Interventions: Drug: Niraparib; Radiation: Re-irradiation (re-RT)

INTERVENTIONS:
Drug: Niraparib — 100 mg, 200 mg, or 300mg oral niraparib once daily.
  Other Names: Zejula
Radiation: Re-irradiation (re-RT) — Intensity modulated radiotherapy (IMRT)-based re-RT for a total dose of 35 Gy in 10 daily fractions.

SUMMARY:
The goal of this clinical trial is to investigate a drug called niraparib in patients with glioblastoma that was previously treated but has returned (called recurrent glioblastoma, or rGBM).

Through this study, investigators would like to find out the best dose of niraparib to give to treat the disease when given together with radiotherapy (known in this study as reirradiation, or re-RT).

Patients receive 10 doses of reirradiation over approximately 2 weeks. At the same time, niraparib capsules are taken orally at home, every day. Niraparib treatment continues until the patient is required to stop either because the treatment stops working or because of side-effects.

Participants will come into clinic weekly for blood tests and clinical examinations in the first month of treatment. After this, the assessments will be done monthly.

Once the patient has finished niraparib treatment, the patient will enter follow-up and be seen once a year to see if there are any late side-effects from trial treatment, how the disease is doing, and if further treatments have been received for it. This follow-up continues until the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Local recurrence of GBM which can be resected or which is not amenable for surgical resection. Patients who have had surgery may also be included if there is residual enhancing disease on the immediate post-operative MRI or if enhancing disease develops on subsequent follow-up imaging
* Recurrent tumour visible on MRI-T1-Gd with the diameter measuring ≤6cm
* Prior history of standard dose, conventionally fractionated CNS radiotherapy (i.e. 54-60Gy in 28-33 fractions)
* At least 6 months since the end of pre-irradiation
* < 2 prior lines of chemotherapy
* Karnofsky Performance Score (KPS) ≥ 70%
* Age ≥ 18 years
* Written informed consent
* Adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1.5x109/L
  * platelets ≥ 100 x109/L
  * haemoglobin > 9.0 g/dL
  * total bilirubin ≤ 1.5 x upper limit of normal (ULN) (≤2.0 in patients with known Gilbert's syndrome) OR direct bilirubin ≤ 1 x ULN
  * Aspartate or alanine transferase (AST or ALT) ≤2.5 x ULN
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
* Negative serum or urine pregnancy test for women of childbearing potential (WOCBP)
* Willing to comply with the contraceptive requirements of the trial (see section 6.3 of protocol for details)
* Patients receiving corticosteroids may continue to receive them as long as their dose is stable (i.e. not increased by >2mg) for at least 1-2 weeks prior to initiating protocol therapy
* Agree to not donate blood during trial treatment or for 90 days after the last dose of niraparib
* Normal blood pressure or adequately treated and controlled hypertension

Exclusion Criteria:

* Concurrent participation in another interventional clinical trial
* Tumour progression or recurrence within 3 months of initial concurrent chemoradiation
* Heart failure (compensate or decompensate)
* Previous treatment with PARP inhibitors
* Previous treatment with re-RT
* Women who are pregnant or breast feeding or plan to breastfeed during trial treatment or for 30 days after the last dose of niraparib
* Major surgical procedure within 3 weeks prior to the first dose niraparib. Note: Patient must have recovered from any surgical effects before the first dose of niraparib
* Received any investigational therapy within 4 weeks prior to, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, the first dose of niraparib
* Known hypersensitivity to niraparib components or excipients
* Received a transfusion (platelets or red blood cells) within 4 weeks prior to the first dose of niraparib
* Received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior to the first dose of niraparib
* Known history of Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Known history of a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days of registration) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Prior malignancy (known diagnosis, detection, or treatment of another type of cancer) within 2 years prior to the first dose of niraparib (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated)
* Known leptomeningeal disease, multifocal GBM, or radiologic signs of CNS hemorrhage
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected) infections
* Live vaccines within 30 days prior to the first dose of niraparib while participating in this clinical study
* If being considered for 300mg dose only:
* patient weight <77Kg
* platelet count of <150 x 109/L
* Patient is immunocompromised. Patients with splenectomy are not excluded. Patients with known human immunodeficiency virus (HIV) are not excluded if they meet the following criteria:
* Cluster of differentiation 4 (CD4) ≥350/μL and viral load <400 copies/mL
* No history of acquired immunodeficiency syndrome-defining opportunistic infections within 12 months prior to enrolment.
* No history of HIV-associated malignancy for the past 5 years.
* Concurrent antiretroviral therapy as per the most current National Institutes of Health (NIH) Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents Living with HIV [NIH, 2021] started <4 weeks prior to study enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) as assessed by CTCAE v5.0 | DLTs with an onset date within the first cycle of treatment (typically 28 days) will be assessed.
  DLTs will be assessed in order to determine the maximum tolerated dose of niraparib given concurrently with re-RT.

SECONDARY OUTCOMES:
Safety and tolerability of niraparib given concurrently with re-RT. | Adverse events will be reported until 30 calendar days post last niraparib and/or post last investigational treatment (re-RT) administration.
  Safety and tolerability of niraparib given concurrently with re-RT, characterised in terms of adverse events as assessed by CTCAE v5.0.
Overall survival (OS) | From trial treatment start date until date of death, assessed at 9 months
  Death
Progression-free survival (PFS) | From trial treatment start date until disease progression or death, whichever occurs first, assessed up to 9 months.
  Disease progression or death
Best Overall Objective Response Rate | From trial treatment start date through to end of trial, assessed at 12 months
  Frequency and percentage of patients who experienced a Complete Response (CR), Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD)
Time to treatment failure (TTF) | From trial treatment start date until early treatment discontinuation, progression, starting further treatment or death, whichever occurs first assessed up to 9 months.
  Treatment failure classified as early treatment discontinuation, progression, starting further treatment or death.
Duration on Treatment | From trial treatment start date until treatment discontinuation, assessed at 12 months
  Median time on trial treatment will be presented.
Treatment Compliance | From trial treatment start date until treatment discontinuation, assessed at 12 months
  Reasons for treatment delays, dose omissions, dose reductions and treatment discontinuation.
Health-related Quality of life (HRQoL): QLQ-C30 | From screening up to 9 months, at specific time points
  HRQoL assessed by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30, scored according to EORTC manual guideline. Score range is 0-100, with 100 being the highest response level.
Health-related Quality of life (HRQoL): QLQ-BN20 | From screening up to 9 months, at specific time points
  HRQoL assessed by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-BN20, scored according to EORTC manual guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Dusan Milanovic, Principal Investigator — The Christie NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cancer Research UK & UCL Cancer Trials Centre — http://www.ctc.ucl.ac.uk/